CLINICAL TRIAL: NCT04838366
Title: The Effect of Pre-operative Carbohydrate Loading in Femur Fracture: A Randomized Controlled Trial
Brief Title: Effect of Preoperative Carbohydrate Loading in Femur Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Police Force Hospital, Nepal (Other Government)
Responsible Party: Principal Investigator, Dev Ram Sunuwar, Dietitian/Researcher, Armed Police Force Hospital, Nepal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Carbohydrateloading
Record Dates: First submitted 2021-04-03; First posted 2021-04-09 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2021-04

CONDITIONS: Femur Fracture
Keywords: Femur fracture; Carbohydrate loading; Visual Analogue Score (VAS); Cumulative Ambulatory Score (CAS)
MeSH Terms: conditions — Femoral Fractures | interventions — Diet, Carbohydrate Loading

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio, and assigned into study group and control group randomly through computer generated block randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The study group will be intervened with carbohydrate loading as the protocol made by ERAS(Li et al., 2021). We will provide glucose-D.
  Interventions: Dietary Supplement: Carbohydrate loading
- Usual care (No Intervention): The control group will be kept in fasting condition from midnight as a traditional practice in existence.

INTERVENTIONS:
Dietary Supplement: Carbohydrate loading — study group will be intervened with carbohydrate loading as the protocol made by ERAS(Li et al., 2021). Surgical patients will be asked to drink a beverage containing 100 grams carbohydrate the night before surgery. On the day of surgery, patients will drink a beverage containing 50 grams carbohydrate 2 hours before surgery under the supervision of research team member. We will provide glucose-D (Dabur Nepal Private Limited, Bara, Nepal, (Regd No.: 3506/045/046, DFTQC No.: 01-33-55-03-218).
  Arms: Intervention

SUMMARY:
Femur fracture is very common in older people. It makes the people bedridden for long time at hospital. The fracture of femur is generally managed by the surgical procedure. Prolonged fasting for surgery makes the patients harassed physically as well as mentally. The long fasting state emphasizes the body more in catabolic state which increases the insulin resistivity. Pre-operative carbohydrate loading before two hours the surgery has been launched in practice to overcome these problems in the world context, however it is not in existence in Nepal. The aim of the study is to evaluate the effect of pre-operative carbohydrate loading in the case of femur fracture surgery.

This study utilize a hospital based randomized control trial study design to assess the effect of carbohydrate loading before two hours the surgery over the completely fasting state. A representative sample size of 66 patients (control group =33 and study group =33) aged 50 years and above having femur fracture planned for surgery will be selected for research. The pre-operative nutritional status will be identified and the post-operative outcomes will be measured by Visual Analogue Score (VAS) and Cumulative Ambulatory Score (CAS). Statistical analysis will be performed using chi square test, independent sample t-test or Mann-Whitney U test to compare between the outcome of study groups and control groups. The outcome of the study may provide a platform to the anaesthesiologists and surgeons towards the emerging concept of pre-operative carbohydrate loading practice in Orthopedics surgery in Nepal.

DETAILED DESCRIPTION:
Femur fracture is one of the most common cause for hospital stay in the case of elder people. Besides these, the patients have the stress of surgery. According to existing practice, the patients are kept in fasting state from the midnight that makes the patients physically as well as mentally discomfort. The patients go in the catabolic state. In addition to these, the prevalence of malnutrition in older people having hip fracture ranges from 2% to 63%. Now the new concept has been launched that the patients should be fed 50 gram carbohydrate two hours prior to the surgery, called carbohydrate loading. The study reveals that preoperative carbohydrate loading decreases the insulin resistance and improves metabolic functions. It presents the patients in anabolic state rather than catabolic state, resulting in the less post-operative protein and nitrogen loss, which facilitates the wound healing. It improves the recovery rate, and hence decreases the length of post-operative stay at hospital, that brings the smile in the face of patients and reduces the treatment cost too. Similarly, it is also associated with significantly better well-being. In Nepal, there is the practice of giving anesthesia to the patient in complete fasting state.

The prolonged fasting state adds the harassment in the patients. Now, the practice of preoperative carbohydrate loading before two hours of surgery is preferred in the world context to minimize the problem of patients discomfort and to maximize better outcome. However, this type of trend is not practiced in Nepal. Furthermore, the issue of nutrition is not prioritized in orthopedics in Nepal. So, this study will also evaluate the nutritional status of the patients under study to relate with the outcomes.

The sample size will be calculated based on the previous similar study with a Mean + SE of Cumulative Ambulatory score (Study groups Vs Control groups: 12.76 + 0.33 Vs 12.02 + 0.32). Considering this data with taking α level of significance at 5% and power of 80%, the sample size will be calculated using test comparing independent two means in Stata/MP version 14.1 (StataCorp LP, College Station, Texas). The calculated sample size is 60. To take into account with 10% loss through follow-up and drop out, the total sample size will be 66 (33 participants in each group.)

ELIGIBILITY:
Inclusion Criteria:

* • Patients of age 50 years and above with femur fracture scheduled for surgery under spinal anesthesia

Exclusion Criteria:

* Pre-existing diabetes (Type I or II)
* Previous intolerance to carbohydrate drinks
* Pathological fracture or any suspected pathology
* Failure case of surgery or non-union case

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
wellbeing of the patients | One week
  The visual analog scale (VAS) will be used to evaluate the well-being of the patients (pain, thirst, and hungry) after surgery. The VAS scores will be recorded on the morning of the first and second postoperative day (24, and 48 hours post-operative, respectively) for groups.
Functional mobility of the patients | One week
  The Cumulative Ambulatory Score (CAS) will be applied to find out the mobility function after surgery. The CAS scores will be recorded on the morning of the first, second, and third postoperative day (24, 48, and 72 hours post-operative, respectively) for both groups.

SECONDARY OUTCOMES:
Change serum albumin level | One week
  Serum albumin level will be assessed after surgery for both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Dev Ram Sunuwar, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bilku DK, Dennison AR, Hall TC, Metcalfe MS, Garcea G. Role of preoperative carbohydrate loading: a systematic review. Ann R Coll Surg Engl. 2014 Jan;96(1):15-22. doi: 10.1308/003588414X13824511650614. PMID 24417824
- [Result] Breedveld-Peters JJ, Reijven PL, Wyers CE, van Helden S, Arts JJ, Meesters B, Prins MH, van der Weijden T, Dagnelie PC. Integrated nutritional intervention in the elderly after hip fracture. A process evaluation. Clin Nutr. 2012 Apr;31(2):199-205. doi: 10.1016/j.clnu.2011.10.004. Epub 2011 Oct 28. PMID 22035956
- [Result] Li ZE, Lu SB, Kong C, Sun WZ, Wang P, Zhang ST. Comparative short-term outcomes of enhanced recovery after surgery (ERAS) program and non-ERAS traditional care in elderly patients undergoing lumbar arthrodesis: a retrospective study. BMC Musculoskelet Disord. 2021 Mar 17;22(1):283. doi: 10.1186/s12891-021-04166-z. PMID 33731057
- [Result] From the American Association of Neurological Surgeons (AANS), American Society of Neuroradiology (ASNR), Cardiovascular and Interventional Radiology Society of Europe (CIRSE), Canadian Interventional Radiology Association (CIRA), Congress of Neurological Surgeons (CNS), European Society of Minimally Invasive Neurological Therapy (ESMINT), European Society of Neuroradiology (ESNR), European Stroke Organization (ESO), Society for Cardiovascular Angiography and Interventions (SCAI), Society of Interventional Radiology (SIR), Society of NeuroInterventional Surgery (SNIS), and World Stroke Organization (WSO); Sacks D, Baxter B, Campbell BCV, Carpenter JS, Cognard C, Dippel D, Eesa M, Fischer U, Hausegger K, Hirsch JA, Shazam Hussain M, Jansen O, Jayaraman MV, Khalessi AA, Kluck BW, Lavine S, Meyers PM, Ramee S, Rufenacht DA, Schirmer CM, Vorwerk D. Multisociety Consensus Quality Improvement Revised Consensus Statement for Endovascular Therapy of Acute Ischemic Stroke. Int J Stroke. 2018 Aug;13(6):612-632. doi: 10.1177/1747493018778713. Epub 2018 May 22. No abstract available. PMID 29786478
- [Derived] Chaudhary NK, Sunuwar DR, Sharma R, Karki M, Timilsena MN, Gurung A, Badgami S, Singh DR, Karki P, Bhandari KK, Pradhan PMS. The effect of pre-operative carbohydrate loading in femur fracture: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Aug 30;23(1):819. doi: 10.1186/s12891-022-05766-z. PMID 36042436
- See also: Chada, R. R., Maryada, V. R., Mulpur, P., Reddy, A., & Maska, A. (2019). Does Preoperative Carbohydrate Loading Help Outcomes in Total Knee Replacement Surgery? J Nutri Med Diet Care, 5(1), 36. — https://clinmedjournals.org/articles/jnmdc/journal-of-nutritional-medicine-and-diet-care-jnmdc-5-036.pdf